CLINICAL TRIAL: NCT03135899
Title: A Two Part Phase I, Multiple-dose, Single- and Double-blind, Randomised, Double-dummy, Placebo-controlled, Four-way Crossover Study to Assess Safety and Tolerability of BI 443651 Via Respimat® Versus Placebo Via Respimat® in Subjects With Mild Asthma Following Methacholine Challenge.
Brief Title: BI 443651 Methacholine Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1363.7; 2016-001506-42 (EudraCT Number)
Record Dates: First submitted 2017-04-26; First posted 2017-05-02 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 443651 (Experimental)
  Interventions: Drug: BI 443651
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 443651 — Three doses, each 12 hours apart
  Arms: BI 443651
Drug: Placebo — Three doses, each 12 hours apart
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate safety and tolerability of three consecutive administrations, 12 hours apart, at three different dose-levels of BI 443651 administered via oral inhalation in male and female mild asthmatic subjects after a bolus methacholine challenge.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects must have a diagnosis of asthma by a physician at least 3 months prior to screening. The diagnosis of asthma must meet the following spirometric criteria:

  -- Pre-bronchodilator clinic measured FEV1 >=70% of predicted normal (calculated by the Global Lung Function Initiative equation (GLI)) measured >= 8 hours after the last use of short acting bronchodilator at the screening visit and on the day of randomisation.
* Age >= 18 <= 60 years. Subjects must be within the eligible age range on the day of signing informed consent.
* Diagnosis of asthma must have been made before the subject's age of 40. Or If the subject is >= 40 years and the diagnosis has not yet been recorded in the subject's medical files, the investigator should assess whether the subject's medical history (e.g. symptoms and prescribed medications) confirms the subject suffered from asthma since before the age of 40. If so, this subject may be considered for inclusion after consultation with the sponsor.
* ACQ value < 1.5 at the screening visit.
* PD20 (Provocative dose causing at least a 20% decline in FEV1) at the screening visit of methacholine <= 1mg
* Body mass index (BMI) >= 18.5 and <= 32.0 kg/m2 at the screening visit
* Subjects must be able to perform all study related procedures and assessments, including pulmonary function tests, as required by the protocol.

Exclusion criteria:

* Significant pulmonary diseases other than asthma (up to GINA treatment step 2) or other medical conditions (as determined by medical history, examination and clinical investigations at screening) that may, in the opinion of the investigator result in any of the following:

  * Put the subject at risk because of participation in the study
  * Influence the results of the study
  * Cause concern regarding the subject's ability to participate in the study.
* Respiratory tract infection or asthma exacerbation in the 4 weeks prior to the screening visit. Subjects can be rescreened 4 weeks after resolution of the infection or exacerbation.
* Hospitalisation for asthma exacerbation within 3 months or intubation for asthma within 3 years of the screening visit.
* Serum potassium measurement above the ULN at the screening visit. Any value about the ULN excludes the subject irrespective of clinical relevance.
* Blood donation (more than 100mL within 30 days prior to the administration of trial medication or intended during the trial)
* Subjects who have been treated with any of the following asthma medications in the given interval prior to Visit 1:

  * Non-approved asthma therapies such as methotrexate,
  * Intravenous, intramuscular or oral corticosteroids
  * Inhaled corticosteroids (iCS) other than low dose iCS (defined as equivalent to equal to, or less than 250 μg fluticasone / day)
  * A long acting beta agonist or anticholinergic bronchodilator (Visit 1), including fixed dose beta agonist/inhaled corticosteroid combinations and oral bronchodilators.
  * A biological based antagonist therapy including Omalizumab, or immune modulators
  * Asthma controller medications (e.g: leukotriene modifier, methylxanthines, nedocromil or cromolyn sodium)
  * Mucolytics
  * Systemically available immunomodulatory treatments for allergic rhinitis or atopic dermatitis.
* Use of any diuretics (including loop diuretics or potassium sparing diuretics (such as amiloride), renin-angiotensin antihypertensive drugs in the 28 days prior to the screening visit (Visit 1)
* Use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval within 10 days prior to the randomisation visit.
* A marked baseline prolongation of QT/QTcF interval (such as QTcF intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening and prior to randomisation
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* History of relevant allergies/hypersensitivities (including allergy to the trial medication or its excipients)
* Contraceptive measures for male and female patients may be required
* Current smokers or ex-smokers who have given up smoking for < 12 months and / or have a smoking pack history of > 5 pack years (1 pack year = 20 cigarettes per day for 1 year of 5 cigarettes per day for 4 years)
* Further exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- The Medicines Evaluation Unit, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with mild asthma were recruited in this trial, which was split into 2 parts. Part 1 was a multiple-dose, single-blind, double-dummy, randomized, 4-way crossover trial with dose ordered sequences. Part 2 was a multiple-dose, double-blind, double-dummy, randomized, 4-way crossover trial.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist site which ensured that they (the patients) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Placebo/BI 443651 100/400/1200 Micro Gram (μg) - Part 1: Patients were orally administered placebo matched to BI 443651 inhalation solution in period 1, followed by BI 443651 100 micro gram (μg) inhalation solution in period 2, BI 443651 400 μg inhalation solution in period 3 and BI 443651 1200 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 100 μg/Placebo/BI 443651 400/1200 μg - Part 1: Patients were orally administered BI 443651 100 μg inhalation solution in period 1, followed by placebo matched to BI 443651 inhalation solution in period 2, BI 443651 400 μg inhalation solution in period 3 and BI 443651 1200 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 100/400 μg/Placebo/BI 443651 1200 μg - Part 1: Patients were orally administered BI 443651 100 μg inhalation solution in period 1, followed by BI 443651 400 μg inhalation solution in period 2, placebo matched to BI 443651 inhalation solution in period 3 and BI 443651 1200 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 100/400/1200 μg/Placebo - Part 1: Patients were orally administered BI 443651 100 μg inhalation solution in period 1, followed by BI 443651 400 μg inhalation solution in period 2, BI 443651 1200 μg inhalation solution in period 3 and placebo matched to BI 443651 inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- Placebo/BI 443651 100/400/1200 μg - Part 2: Patients were orally administered placebo matched to BI 443651 inhalation solution in period 1, followed by BI 443651 100 μg inhalation solution in period 2, BI 443651 400 μg inhalation solution in period 3 and BI 443651 1200 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 400/1200 μg/Placebo/BI 443651 100 μg - Part 2: Patients were orally administered BI 443651 400 μg inhalation solution in period 1, followed by BI 443651 1200 μg inhalation solution in period 2, placebo matched to BI 443651 inhalation solution in period 3 and BI 443651 100 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 100 μg/Placebo/BI 443651 1200/400 μg - Part 2: Patients were orally administered BI 443651 100 μg inhalation solution in period 1, followed by placebo matched to BI 443651 inhalation solution in period 2, BI 443651 1200 μg inhalation solution in period 3 and BI 443651 400 μg inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
- BI 443651 1200/400/100 μg/Placebo - Part 2: Patients were orally administered BI 443651 1200 μg inhalation solution in period 1, followed by BI 443651 400 μg inhalation solution in period 2, BI 443651 100 μg inhalation solution in period 3 and placebo matched to BI 443651 inhalation solution in period 4, each treatment was administered via Respimat® inhaler. All treatment periods were separated by a washout period of 14-28 days.
Period: Overall Study
Arm/Group | Placebo/BI 443651 100/400/1200 Micro Gram (μg) - Part 1 | BI 443651 100 μg/Placebo/BI 443651 400/1200 μg - Part 1 | BI 443651 100/400 μg/Placebo/BI 443651 1200 μg - Part 1 | BI 443651 100/400/1200 μg/Placebo - Part 1 | Placebo/BI 443651 100/400/1200 μg - Part 2 | BI 443651 400/1200 μg/Placebo/BI 443651 100 μg - Part 2 | BI 443651 100 μg/Placebo/BI 443651 1200/400 μg - Part 2 | BI 443651 1200/400/100 μg/Placebo - Part 2
Started | 1 | 1 | 1 | 1 | 8 | 9 | 8 | 8
Completed | 1 | 1 | 1 | 1 | 8 | 7 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Failed spirometry,unable to repeat visit | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all patients who had been randomised and treated with at least 1 dose of trial medication. The treatment assignment was determined based on the first treatment the patients received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/BI 443651 100/400/1200 Micro Gram (μg) - Part 1 | BI 443651 100 μg/Placebo/BI 443651 400/1200 μg - Part 1 | BI 443651 100/400 μg/Placebo/BI 443651 1200 μg - Part 1 | BI 443651 100/400/1200 μg/Placebo - Part 1 | Placebo/BI 443651 100/400/1200 μg - Part 2 | BI 443651 400/1200 μg/Placebo/BI 443651 100 μg - Part 2 | BI 443651 100 μg/Placebo/BI 443651 1200/400 μg - Part 2 | BI 443651 1200/400/100 μg/Placebo - Part 2 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 9 | 8 | 8 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 | 41 | 59 | 35 | 39.1 (10.5) | 36.1 (10.3) | 35.4 (11.1) | 35.9 (11.7) | 37.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Male | 1 | 1 | 1 | 1 | 6 | 8 | 8 | 8 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 8 | 9 | 8 | 8 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  White | 1 | 1 | 1 | 1 | 7 | 9 | 4 | 4 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Maximum Forced Expiratory Volume Within 1 Second (FEV1) Reduction Following Bolus Methacholine Challenge in Part 1
Description: Absolute change from baseline in maximum forced expiratory volume within 1 second (FEV1) reduction following bolus methacholine challenge in Part 1 was defined as the difference between the maximum reduction in FEV1 obtained during the treatment challenge and during the baseline challenge.
Time Frame: Baseline and Day 2
Population: Methacholine set (MCS): The MCS included all patients in the TS who provided at least one pair (baseline and end-of-treatment) of evaluable measures of spirometry parameters that were not excluded due to use of rescue medication within 3 hours (h) after start of bolus methacholine challenge.
Measure: Mean (Standard Deviation); unit: Litres (L)
Groups:
- Placebo - Part 1: Patients were orally administered 4 actuations, thrice 12 hours (h) apart, of placebo matched with BI 443651 inhalation solution via Respimat® inhaler.
- BI 443651 100 μg - Part 1: Patients were orally administered 1 actuation of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 400 μg - Part 1: Patients were orally administered 4 actuations, thrice 12 h apart, of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 1200 μg - Part 1: Patients were orally administered 4 actuations, thrice 12 h apart, of BI 443651 300 μg inhalation solution via Respimat® inhaler.
Arm/Group | Placebo - Part 1 | BI 443651 100 μg - Part 1 | BI 443651 400 μg - Part 1 | BI 443651 1200 μg - Part 1
Number analyzed (Participants) | 4 | 4 | 4 | 4
Litres (L) | 0.018 (0.554) | 0.390 (0.261) | -0.195 (0.431) | 0.272 (0.268)

2. Primary Outcome: Absolute Change From Baseline in Maximum Forced Expiratory Volume Within 1 Second (FEV1) Reduction Following Bolus Methacholine Challenge in Part 2.
Description: Absolute change from baseline in maximum FEV1 reduction following bolus methacholine challenge in Part 2 was defined as the difference between the maximum reduction in FEV1 obtained during the treatment challenge and during the baseline challenge.
Time Frame: Baseline and Day 2
Population: MCS
Measure: Least Squares Mean (Standard Error); unit: Litres (L)
Groups:
- Placebo - Part 2: Patients were orally administered 4 actuations, thrice 12 hours (h) apart, of placebo matched with BI 443651 inhalation solution via Respimat® inhaler.
- BI 443651 100 μg - Part 2: Patients were orally administered 1 actuation of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 400 μg - Part 2: Patients were orally administered 4 actuations, thrice 12 h apart, of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 1200 μg - Part 2: Patients were orally administered 4 actuations, thrice 12 h apart, of BI 443651 300 μg inhalation solution via Respimat® inhaler.
Arm/Group | Placebo - Part 2 | BI 443651 100 μg - Part 2 | BI 443651 400 μg - Part 2 | BI 443651 1200 μg - Part 2
Number analyzed (Participants) | 31 | 31 | 32 | 31
Litres (L) | 0.005 (0.056) | 0.064 (0.056) | -0.032 (0.055) | -0.152 (0.056)
Statistical Analysis 1: Comparison: Placebo - Part 2 vs BI 443651 100 μg - Part 2; The mixed effects model included 'treatment' and 'period' as fixed effects, 'patient' as a random effect, and 'period baseline' as well as 'patient baseline' as covariates. No hypothesis was tested. The patient baseline was obtained by calculating the mean of the period baselines for each patient. Covariance structure variance component (VC) was used for random subject effect; Test type: Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 90% CI 2-sided [-0.048 to 0.165], Standard Error of Mean 0.064 — BI 443651 100 μg is compared to placebo
Statistical Analysis 2: Comparison: Placebo - Part 2 vs BI 443651 400 μg - Part 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.037, 90% CI 2-sided [-0.144 to 0.070], Standard Error of Mean 0.064 — BI 443651 400 μg is compared to placebo
Statistical Analysis 3: Comparison: Placebo - Part 2 vs BI 443651 1200 μg - Part 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.157, 90% CI 2-sided [-0.266 to -0.047], Standard Error of Mean 0.066 — BI 443651 1200 μg is compared to placebo

3. Secondary Outcome: Relative Change From Baseline in FEV1 Area Under the Curve Over the Time Interval From 0 to Timepoint tz (FEV1 AUC0-tz) Following Bolus Methacholine Challenge in Part 1
Description: Relative change from baseline in FEV1 area under the curve over the time interval from 0 to timepoint tz (FEV1 AUC0-tz) following bolus methacholine challenge in Part 1 was defined as the ratio of FEV1 AUC0-tz obtained during the treatment challenge and during the baseline challenge, where the time tz refers to the last time point before recovery of FEV1 to within 95% of post-diluent value.
Time Frame: Baseline and Day 2
Population: MCS
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo - Part 1 | BI 443651 100 μg - Part 1 | BI 443651 400 μg - Part 1 | BI 443651 1200 μg - Part 1
Number analyzed (Participants) | 4 | 4 | 4 | 4
Ratio | 1.097 (0.849) | 0.625 (0.262) | 0.925 (0.364) | 0.296 (0.218)

4. Secondary Outcome: Relative Change From Baseline in FEV1 Area Under the Curve Over the Time Interval From 0 to Timepoint tz (FEV1 AUC0-tz) Following Bolus Methacholine Challenge in Part 2
Description: Relative change from baseline in FEV1 area under the curve over the time interval from 0 to timepoint tz (FEV1 AUC0-tz) following bolus methacholine challenge in Part 2 was defined as the ratio of FEV1 AUC0-tz obtained during the treatment challenge and during the baseline challenge, where the time tz refers to the last time point before recovery of FEV1 to within 95% of post-diluent value. Geometric mean is actually adjusted geometric mean. Standard error presented here is a geometric standard error.
Time Frame: Baseline and Day 2
Population: MCS
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Placebo - Part 2 | BI 443651 100 μg - Part 2 | BI 443651 400 μg - Part 2 | BI 443651 1200 μg - Part 2
Number analyzed (Participants) | 31 | 31 | 32 | 31
Ratio | 0.863 (1.152) | 0.665 (1.152) | 0.799 (1.150) | 0.729 (1.152)
Statistical Analysis 1: Comparison: Placebo - Part 2 vs BI 443651 100 μg - Part 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio = 0.770, 90% CI 2-sided [0.595 to 0.977], Standard Error of Mean 1.168 — BI 443651 100 μg is compared to placebo. Standard error of the mean is actually geometric standard error
Statistical Analysis 2: Comparison: Placebo - Part 2 vs BI 443651 400 μg - Part 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio = 0.926, 90% CI 2-sided [0.715 to 1.199], Standard Error of Mean 1.168 — BI 443651 400 μg is compared to placebo. Standard error of the mean is actually geometric standard error
Statistical Analysis 3: Comparison: Placebo - Part 2 vs BI 443651 1200 μg - Part 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Mixed Models Analysis; Geometric Mean Ratio = 0.845, 90% CI 2-sided [0.651 to 1.095], Standard Error of Mean 1.169 — BI 443651 1200 μg is compared to placebo. Standard error of the mean is actually geometric standard error

5. Secondary Outcome: Time to Recovery of FEV1 to Within 95% of Post-diluent Value in Part 1
Description: Time to recovery of FEV1 to within 95% of post-diluent value in Part 1 was defined as the time from maximum reduction to last time before recovery to within 95% of the value obtained pre-methacholine challenge during the respective challenge.
Time Frame: Day 2
Population: MCS
Measure: Median (Inter-Quartile Range); unit: hours (h)
Arm/Group | Placebo - Part 1 | BI 443651 100 μg - Part 1 | BI 443651 400 μg - Part 1 | BI 443651 1200 μg - Part 1
Number analyzed (Participants) | 4 | 4 | 4 | 4
hours (h) | 0.775 [0.283 to 2.752] | 0.452 [0.217 to 1.185] | 0.751 [0.311 to 2.336] | 0.597 [0.266 to 0.996]

6. Secondary Outcome: Time to Recovery of FEV1 to Within 95% of Post-diluent Value in Part 2
Description: Time to recovery of FEV1 to within 95% of post-diluent value in Part 2 was defined as the time from maximum reduction to last time before recovery to within 95% of the value obtained pre-methacholine challenge during the respective challenge. Median is actually model-based median.
Time Frame: Day 2
Population: MCS
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Placebo - Part 2 | BI 443651 100 μg - Part 2 | BI 443651 400 μg - Part 2 | BI 443651 1200 μg - Part 2
Number analyzed (Participants) | 31 | 31 | 32 | 31
h | 0.65 [0.33 to 0.74] | 0.48 [0.30 to 0.52] | 0.44 [0.30 to 0.48] | 0.32 [0.16 to 0.48]
Statistical Analysis 1: Comparison: Placebo - Part 2 vs BI 443651 100 μg - Part 2; The cox proportional hazard model included treatment and period as fixed effect and patient baseline as covariate. No hypothesis was tested. The patient baseline was obtained by calculating the median of the period baselines for each patient. A hazard ratio greater than 1 gives that active treatment is not-inferior to placebo; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 2.27, 95% CI 2-sided [1.31 to 3.95] — BI 443651 100 μg is compared to placebo
Statistical Analysis 2: Comparison: Placebo - Part 2 vs BI 443651 400 μg - Part 2; [analysis description as in outcome 6, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 2.08, 95% CI 2-sided [1.22 to 3.53] — BI 443651 400 μg is compared to placebo
Statistical Analysis 3: Comparison: Placebo - Part 2 vs BI 443651 1200 μg - Part 2; [analysis description as in outcome 6, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 2.59, 95% CI 2-sided [1.50 to 4.47] — BI 443651 1200 μg is compared to placebo

ADVERSE EVENTS:
Time Frame: From the first drug administration until 14 days after the last drug administration, up to 16 days.
Description: Treated set (TS): The TS included all patients who had been randomised and treated with at least 1 dose of trial medication. The treatment assignment was determined based on the first treatment the patients received.
Groups:
- Placebo - Part 1 & Part 2: Patients were orally administered 4 actuations of placebo matched with BI 443651 inhalation solution via Respimat® inhaler.
- BI 443651 100 Microgram (μg) - Part 1 & Part 2: Patients were orally administered 1 actuation of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 400 μg - Part 1 & Part 2: Patients were orally administered 4 actuations of BI 443651 100 μg inhalation solution via Respimat® inhaler.
- BI 443651 1200 μg - Part 1 & Part 2: Patients were orally administered 4 actuations of BI 443651 300 μg inhalation solution via Respimat® inhaler.
Arm/Group | Placebo - Part 1 & Part 2 | BI 443651 100 Microgram (μg) - Part 1 & Part 2 | BI 443651 400 μg - Part 1 & Part 2 | BI 443651 1200 μg - Part 1 & Part 2
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 9/35 | 21/35 | 24/36 | 26/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Part 1 & Part 2 (N=35) | BI 443651 100 Microgram (μg) - Part 1 & Part 2 (N=35) | BI 443651 400 μg - Part 1 & Part 2 (N=36) | BI 443651 1200 μg - Part 1 & Part 2 (N=36)
Chest discomfort (General disorders) | 0 | 0 | 2 | 11
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 5 | 12 | 15
Headache (Nervous system disorders) | 6 | 7 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03135899/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03135899/SAP_001.pdf